CLINICAL TRIAL: NCT02331329
Title: Evaluation of NICOM (Bioreactance) for the Non-invasive Determination of Cardiac Output
Status: Completed | Type: Observational
Sponsor: Universitätsmedizin Mannheim (Other)
Responsible Party: Principal Investigator, Joachim Saur, senior physician, Universitätsmedizin Mannheim
Other Study IDs: NICOM
Record Dates: First submitted 2015-01-02; First posted 2015-01-06 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2015-01

CONDITIONS: Cardiac Disease
Keywords: Accuracy of NICOM; precision of NICOM
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: NICOM cardiac output measurement
Device: Cardiac MRT cardiac output measurement

SUMMARY:
Cardiac output (CO) is an important parameter in the diagnosis and therapy of cardiac diseases. The current standard methods for the determination of CO, however, are either invasive (e.g. right heart catheterization) or technically expendable and expensive (magnetic resonance tomography, MRT). Therefore, the aim of the study at hand was to evaluate NICOM (bioreactance) as a new method for determinion of CO and to compare this new technique to MRT.

ELIGIBILITY:
Inclusion Criteria:

* indication for cardiac magnetic resonance imaging

Exclusion Criteria:

* pace maker
* patient unwilling to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hemodynamically and respiratory stable patients undergoing cardiac magnetic resonance imaging with a clinical indication
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2013-07; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
agreement of NICOM and MRT cardiac output measurements | at time of inclusion
precision of NICOM cardiac output measurements | at time of inclusion